CLINICAL TRIAL: NCT07403227
Title: Comparative Effects of Muscle Energy Technique and Modified Active Release Technique in Patients With Scapulocostal Syndrome.
Brief Title: Comparative Effects of Muscle Energy Technique and Modified Active Release Technique in Scapulocostal Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/01105
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Scapulocostal Syndrome
Keywords: Chronic Neck Pain; Muscle Energy Technique; Myofascial Release Therapy; Neck Ache; Neck Disability; Manual Therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental)
  Interventions: Other: Muscle Energy Technique; Other: Conventional Physical Therapy
- Modified Active Release Technique (Active Comparator)
  Interventions: Other: Modified Active Release Technique; Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Muscle Energy Technique — Muscle Energy Technique (PIR) began by putting the muscles in stretched position. An isometric contraction was exerted against minimum resistance. Followed by Relaxation, then gentle stretch followed as the muscle releases. Tight, tender muscles commonly suffering with pain undergoes such techniques. All the contraction were hold for 10 seconds for each muscle i.e. 10 repetitions followed with 20 seconds rest time.
  1. MET for upper Trapezius Muscle.
  2. MET for Levator scapulae Muscle
  3. MET for Rhomboid muscle
  Other Names: MET
  Arms: Muscle Energy Technique
Other: Modified Active Release Technique — Modified Active Release Technique combined the active movement by patients with the passive movements done by the therapist. During this, participants were instructed to hold every movement for 6seconds with 10 repetitions. Pin and stretch type of modified active release technique was used in the study.
  1. Modified Active Release Technique for Upper trapezius:
  2. Modified Active Release Technique for Levator Scapulae:
  3. Modified Active Release Technique for Rhombhoids.
  Other Names: mART
  Arms: Modified Active Release Technique
Other: Conventional Physical Therapy — * Hot pack for 10 minutes.
  * Transcutaneous electrical nerve stimulation (TENS) (frequency: 2Hz and pulse duration 200 μs, 10 minutes
  Other Names: Baseline Treatment

SUMMARY:
The study was conducted to determine the comparative effects of Muscle Energy Technique and Modified Active Release Technique on Pain, Chest expansion and Functional disability in patients with Scapulocostal Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 yrs.
* Both male and females with shoulder-neck pain.
* NPRS value> than 3.
* Chest expansion value < than 3cm are included.
* Subjects with Upper Trapezius, Levator Scapulae and Rhomboid muscles tenderness.
* Pain duration should be present for at least for 3 months before inclusion in the study.
* Presence of 1 to 3 trigger points in upper trapezius, levator scapulae, and rhombhoids (MTrP) causing referred pain pattern with palpable taut band of muscle.

Exclusion Criteria:

* Thoracic outlet syndrome.
* Brachial neuralgia.
* Local neck and shoulder disorder.
* Adhesive Capsulitis.
* Cervical Radiculopathy.
* Trauma or Injury around Scapular area.
* Past Surgical Area.
* Any cardiovascular or Respiratory pathology.
* People with psychiatric illness such as depression.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | From enrollment to the end of treament at 6 weeks.
  Patient's pain level was accessed using NPRS. It is a tool used to check the severity of pain, on a scale of 0 to 10, 0 indicates no pain, 1-3 means mild pain,4to 6 indicates moderate pain, and 7 to 10 value shows severe pain. Patient rates their level of pain at that time and the less and severe pain level in previous 24 hours, Then the average is taken by using 3 values. Validity of NPRS is 0.86 and reliability 0.96.
Neck Disability Index. | From enrollment to the end of treatment at 6 weeks
  Neck Disability index is a tool to check the neck complaints. Developed from Oswestry Index of neck pain and neck disability index. It is based on activites of daily life and provide a good functional value. This scale consists of 10 sections, each section contains 5 further questions of daily life activities affected, each section scored 0 to 5. The subject was asked to answer these questions. By dividing the total scores over number of questions answered and multiply by 100, the index was calculated. The validity and realibility of NDI is good
Measuring Inches Tape | From enrollment to the end of study at 6 weeks
  Measuring Tape is used to measure Chest expansion. It is a reliable, non-invasive and simple method. Chest Expansion is measured by thoracic girth difference, after maximal inspiration, and at maximal expiration end point. There are several anatomical landmarks to measures upper and lower chest expansion. Anatomical landmarks are 4th intercostal space, axillary lines, and thoracic vertebrae (3rd ,5th .12th) and 10th thoracic vertebrae and xiphoid process. 4th Intercostal space and axillary lines were used to measure chest expansion in this study at both levels. The 2-instruction evaluated were, "breathe in maximally, breathe out maximally". And value were recorded at end of Maximal inhalation and maximal exhalation. A difference in these values were then calculated. An acceptable Reliability by ICC was determined. Value > 0.85 and SEMs < 5%.

SECONDARY OUTCOMES:
ROM Cervical Spine (Flexion) | from enrollment to the end at 6th week of treatment.
  Changes in cervical spine flexion ROM at baseline and at 6th week of intervention was measured using Goniometer.
ROM Cervical Spine (Extension) | from enrollments to the end of treatment at 6 weeks.
  Changes in cervical spine extension ROM at baseline and at 6th week of intervention was measured using Goniometer.
ROM Cervical Spine (Left Lateral Flexion). | From Enrollment to the end of treatment at 6 weeks
  Changes in cervical spine left lateral flexion ROM at baseline and at 6th week of intervention was measured using Goniometer.
ROM Cervical Spine (Right Lateral Flexion) | From enrollment to the end of treatment at 6 weeks.
  Changes in cervical spine right lateral flexion flexion ROM at baseline and at 6th week of intervention was measured using Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Rafia Mannan, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- AAHAD Hospital Sialkot., Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chatchawan U. Comparative study of the immediate therapeutic effects between modified active release technique and traditional Thai massage on pain alteration in patient with scapulocostal syndrome. DOAJ (DOAJ: Directory of Open Access Journals). 2017.
- [Background] Ali S, Ahmad S, Jalal Y, Shah B. Effectiveness of Stretching Exercises Versus Muscle Energy Techniques in the Management of Upper Cross Syndrome: JRCRS. 2017; 5 (1): 12-16. Journal Riphah College of Rehabilitation Sciences. 2017;5(1):12-6.
- [Background] Mishra D, Prakash RH, Mehta J, Dhaduk A. Comparative study of active release technique and myofascial release technique in treatment of patients with upper trapezius spasm. Journal of Clinical and Diagnostic Research. 2018;12(11):17-20.
- [Background] Ganesh B, Patil P, Rodrigues A. Effect of Muscle Energy Technique on Strength and Range of Motion in Young Swimmers with Sick Scapula Syndrome: A Pre-Post Clinical Trial. Indian Journal of Physiotherapy & Occupational Therapy Print-(ISSN 0973-5666) and Electronic-(ISSN 0973-5674). 2020;14(2):45-9.
- [Background] Allison GT, Nagy BM, Hall T. A randomized clinical trial of manual therapy for cervico-brachial pain syndrome -- a pilot study. Man Ther. 2002 May;7(2):95-102. doi: 10.1054/math.2002.0453. PMID 12151246
- [Background] Risalda P, Phansopkar P, Naqvi WM. Effectiveness of active release technique verses conventional physiotherapy in management of upper cross syndrome. Indian Journal of Forensic Medicine & Toxicology. 2021;15(1):246-50.
- [Background] Seo J, Song C, Shin D. A Single-Center Study Comparing the Effects of Thoracic Spine Manipulation vs Mobility Exercises in 26 Office Workers with Chronic Neck Pain: A Randomized Controlled Clinical Study. Med Sci Monit. 2022 Jul 8;28:e937316. doi: 10.12659/MSM.937316. PMID 35799408
- [Background] Abbas AH, Javaid M, Ali A, Ali Z, Mehmood S, Manzoor S. Comparative Efficacy of Muscle Energy Technique and Myofascial Release Technique in Reducing Pain in Upper Cross Syndrome: A Randomised Clinical Trial. The Healer Journal of Physiotherapy and Rehabilitation Sciences. 2025;5(2):228-34.
- [Background] Mohan V, Dzulkifli NH, Justine M, Haron R, Rathinam C. Intrarater reliability of chest expansion using cloth tape measure technique. Bangladesh journal of medical science. 2012;11(4):307-11.
- [Background] Narulkar R, Welling A, Gurudut P, Kage V. Comparing the efficacy of 3-dimensional release technique and modified active release therapy on pain, scapular position and Craniovertebral angle in IT workers with scapulocostal syndrome: A Randomised Clinical Trial. J Bodyw Mov Ther. 2025 Oct;44:80-90. doi: 10.1016/j.jbmt.2025.05.033. Epub 2025 May 23. PMID 40954664
- [Background] Kanhachon W, Boonprakob Y. Modified-Active Release Therapy in Patients with Scapulocostal Syndrome and Masticatory Myofascial Pain: A Stratified-Randomized Controlled Trial. Int J Environ Res Public Health. 2021 Aug 12;18(16):8533. doi: 10.3390/ijerph18168533. PMID 34444281
- [Background] Zahid A, Gull S, Athar M, Khan IU, Maqbool S, Zahid H. Comparative Effectiveness of Scapular Stabilization Exercises with and Without Deep Breathing on Pain and Chest Expansion in Patients with Scapulocostal Syndrome: Scapular Stabilization with Deep Breathing in SCS. Journal of Health and Rehabilitation Research. 2024;4(3).
- [Background] Deka D, Yaduvanshi P, Mozhi A. EFFECT OF MUSCLE ENERGY TECHNIQUE AND MYOFASCIAL RELEASE IN SCAPULOCOSTAL SYNDROME IN COLLEGIATE YOUNG ADULTS.
- [Background] Buttagat V, Taepa N, Suwannived N, Rattanachan N. Effects of scapular stabilization exercise on pain related parameters in patients with scapulocostal syndrome: A randomized controlled trial. J Bodyw Mov Ther. 2016 Jan;20(1):115-122. doi: 10.1016/j.jbmt.2015.07.036. Epub 2015 Jul 26. PMID 26891646